CLINICAL TRIAL: NCT00094822
Title: Pegfilgrastim Given Same Day as or Day After Carboplatin and Docetaxel in Patients With Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: Pegfilgrastim Given Same Day As or Day After Carboplatin and Docetaxel in Advanced Metastatic Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Other Study IDs: 20030123
Record Dates: First submitted 2004-10-27; First posted 2004-10-27 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2009-02

CONDITIONS: Lung Cancer; Non-Small Cell Lung Cancer
Keywords: Metastatic Cancer; Neulasta®; pegfilgrastim
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Pegfilgrastim
  Interventions: Other: PI Discretion
- PLACEBO
  Interventions: Other: PI Discretion

INTERVENTIONS:
Other: PI Discretion — PI Discretion

SUMMARY:
The purpose of this research study is to evaluate the safety and effectiveness of Neulasta® (pegfilgrastim) in reducing infection when given on the same day versus one day after the completion of chemotherapy (docetaxel and carboplatin) in patients with advanced or metastatic non-small cell lung cancer (NSCLC). This study is considered to be "investigational" because previous studies with Neulasta® used next day dosing and not same day dosing.

ELIGIBILITY:
Eligibility Criteria: - Age 18 years or older - Diagnosis of advanced or metastatic non-small cell lung cancer (NSCLC) - Have not received any prior chemotherapy - Have not received radiation therapy or undergone major surgery within the past 2 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced or Metastatic NSCLC
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2003-07; Primary Completion 2005-12 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
incidence of infection | during treatment

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_11_GCSFSD01_20030123.pdf
- See also: FDA-approved Drug Labeling — http://www.neulasta.com/